CLINICAL TRIAL: NCT06628089
Title: Knowledge, and Practice of Helicobacter Pylori Infection Among Primary Healthcare Physicians in Sohag Governorate
Brief Title: Knowledge, and Practice of Helicobacter Pylori Infection
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Esraa Kamal Abdelzaher, Principal investigator, Sohag University
Other Study IDs: EKAbdelzaher
Record Dates: First submitted 2024-10-01; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: A questionnaire about H. Pylori infection, mode of transmission, Symptoms, treatment will be carried to primary health care physicians and will be asked to answer it
  Interventions: Other: Questionnaire
- 2

INTERVENTIONS:
Other: Questionnaire — A questionnaire for primary healthcare physicians designed to evaluate knowledge about H. Pylori mode of transmission, symptoms, complications and treatment.
  Groups: 1

SUMMARY:
Helicobacter Pylori infection is very common in Our community However, it may be misdiagnosed and treated from the start until the patient present with complications. Therefore, it is essential that primary care physicians have the appropriate knowledge for making adequate decisions and preventing incorrect practices that result in elevated costs and absolutely no health benefits for the population. So this study aims to evaluate the knowledge and practice of primary healthcare physicians at Sohag health care units concerning H. Pylori infection.

DETAILED DESCRIPTION:
The most common cause of chronic gastritis is Helicobacter pylori, which can also cause serious gastroduodenal diseases in some patients. These include gastric cancer, gastric mucosa-associated lymphoid tissue (MALT) lymphoma, and gastric and duodenal peptic ulcer disease (PUD). Strong correlations have been shown between H. pylori and a number of extra-gastric illnesses, including vitamin B12 deficiency, idiopathic thrombocytopenic purpura, and unexplained iron-deficiency anemia. Identifying and eliminating H. pylori in people suffering from these conditions is also advised. Furthermore, neurological disorders, cardiovascular disorders, hepatobiliary disorders and autoimmune disorders may be associated with H. pylori infection. Age, ethnicity, degree of hygiene, and social and economic circumstances are risk factors for H. pylori infection An elevated prevalence of gastrointestinal diseases or symptoms (for example, dyspeptic symptoms) in populations where H. pylori infection is high, implies that a large number of subjects receive primary health care.Therefore, it is essential that primary care physicians have the appropriate knowledge for making adequate decisions and preventing incorrect practices that result in elevated costs and absolutely no health benefits for the population.

Since day-to-day clinical practice demonstrates that many healthcare disciplines surprisingly deal with H. pylori infection in the absence of local guidelines on this matter, there has been no study conducted in Sohag Governate evaluated knowledge, practice and attitude about H. pylori among healthcare physicians as of the time I conducted this survey.

ELIGIBILITY:
Inclusion Criteria:

* physicians at primary healthcare units in Sohag governorate

Exclusion Criteria:

* Nonmedical personnel
* GIT specialists
* physicians at secondary or tertiary healthcare centers

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A questionnaire will be carried to the primary healthcare physicians in Sohag governorate, and they will be asked to answer it .
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
determine the knowledge and practice of primary healthcare physicians at Sohag health care units concerning H. Pylori infection through a written questionnaire and they will be asked to answer it | 6 months
  A questionnaire will be carried to the physicians includes questions about Pylori mode of transmission, symptoms, complications, treatment to assess their knowledge and practice of Pylori infection and correct any wrong management of the disease and decrease the rate of Pylori infection in Shage Governorate

IPD SHARING:
Plan to Share IPD: Undecided